CLINICAL TRIAL: NCT02267343
Title: ONO-4538 Phase III Study A Multicenter, Double-Blind, Randomized Study in Patients With Unresectable Advanced or Recurrent Gastric Cancer
Brief Title: Study of ONO-4538 in Unresectable Advanced or Recurrent Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-4538-12
Record Dates: First submitted 2014-10-09; First posted 2014-10-17 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ONO-4538 Arm (Experimental): ONO-4538 3 mg/kg solution intravenously every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Drug: ONO-4538
- Placebo Arm (Placebo Comparator): Placebo intravenously every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-4538
  Arms: ONO-4538 Arm
Drug: Placebo
  Arms: Placebo Arm

SUMMARY:
The purpose of study is to evaluate the efficacy and safety of ONO-4538 in patients with unresectable advanced or recurrent gastric cancer (including esophagogastric junction cancer) refractory to or intolerant of standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men & women ≥20 years of age
* Unresectable advanced or recurrent gastric cancer (including esophagogastric junction cancer)
* Histologically confirmed adenocarcinoma
* Refractory to or intolerant of standard therapy
* ECOG Performance Status score 0 or 1
* A life expectancy of at least 3 months

Exclusion Criteria:

* Current or past history of severe hypersensitivity to any other antibody products
* Patients with multiple primary cancers
* Patients with any metastasis in the brain or meninx that is symptomatic or requires treatment
* Patients with active, known or suspected autoimmune disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to study completion (estimated time frame: 30 months), every 2 weeks in principle

SECONDARY OUTCOMES:
Progression-free survival | Up to study completion (estimated time frame: 30 months), every 2 weeks in principle
Objective response rate | Up to study completion (estimated time frame: 30 months), every 6 weeks in principle
Duration of response | Up to study completion (estimated time frame: 30 months), every 6 weeks in principle
Safety will be analyzed through the incidence of adverse events, serious adverse events | Continuously throughout study treatment and up to 28 days from last dose
Safety will be analyzed through the incidence of laboratory abnormalities | Continuously throughout study treatment and up to 28 days from last dose

CONTACTS AND LOCATIONS:
Overall Officials: Mitsunobu Tanimoto, Study Director — Ono Pharmaceutical Co. Ltd
Locations (36):
- Japan (27):
  - Aichi Clinical Site, Nagoya, Aichi-ken
  - Aomori Clinical Site, Misawa, Aomori
  - Ehime Clinical Site, Matsuyama, Ehime
  - Hokkaido Clinical Site, Sapporo, Hokkaido
  - Hyogo Clinical Site, Akashi, Hyōgo
  - Hyogo Clinical Site, Kobe, Hyōgo
  - Ishikawa Clinical Site, Kanazawa, Ishikawa-ken
  - Kanagawa Clinical Site, Kawasaki, Kanagawa
  - Kanagawa Clinical Site, Sagamihara, Kanagawa
  - Kanagawa Clinical Site, Yokohama, Kanagawa
  - Nagano Clinical Site, Saku, Nagano
  - Osaka Clinical Site, Sayama, Osaka
  - Osaka Clinical Site, Suita, Osaka
  - Osaka Clinical Site, Takatsuki, Osaka
  - Saitama Clinical Site, Kitaadachi, Saitama
  - Shizuoka Clinical Site, Sunto-gun, Shizuoka
  - Tochigi Clinical Site, Shimotsuke, Tochigi
  - Tokyo Clinical Site, Bunkyo-ku, Tokyo
  - Tokyo Clinical Site, Chuo-ku, Tokyo
  - Tokyo Clinical Site, Koto-ku, Tokyo
  - Tokyo Clinical Site, Shinjuku-ku, Tokyo
  - Chiba Clinical Site, Chiba
  - Fukuoka Clinical Site, Fukuoka
  - Gifu Clinical Site, Gifu
  - Hiroshima Clinical Site, Hiroshima
  - Osaka Clinical Site, Osaka
  - Shizuoka Clinical Site, Shizuoka
- South Korea (4):
  - Busan-si Clinical Site, Busan
  - Daegu Clinical Site, Daegu
  - Gyeonggi-Do Clinical Site, Gyeonggi-do
  - Seoul Clinical Site, Seoul
- Taiwan (5):
  - Kaohsiung Clinical Site, Kaohsiung City
  - Taichung Clinical Site, Taichung
  - Tainan Clinical Site, Tainan
  - Taipei Clinical Site, Taipei
  - Taoyuan Clinical Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang YK, Reck M, Nghiem P, Feng Y, Plautz G, Kim HR, Owonikoko TK, Boku N, Chen LT, Lei M, Chang H, Lin WH, Roy A, Bello A, Sheng J. Assessment of hyperprogression versus the natural course of disease development with nivolumab with or without ipilimumab versus placebo in phase III, randomized, controlled trials. J Immunother Cancer. 2022 Apr;10(4):e004273. doi: 10.1136/jitc-2021-004273. PMID 35383114
- [Derived] Kang YK, Boku N, Satoh T, Ryu MH, Chao Y, Kato K, Chung HC, Chen JS, Muro K, Kang WK, Yeh KH, Yoshikawa T, Oh SC, Bai LY, Tamura T, Lee KW, Hamamoto Y, Kim JG, Chin K, Oh DY, Minashi K, Cho JY, Tsuda M, Chen LT. Nivolumab in patients with advanced gastric or gastro-oesophageal junction cancer refractory to, or intolerant of, at least two previous chemotherapy regimens (ONO-4538-12, ATTRACTION-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Dec 2;390(10111):2461-2471. doi: 10.1016/S0140-6736(17)31827-5. Epub 2017 Oct 6. PMID 28993052